CLINICAL TRIAL: NCT02766309
Title: The Correlation Between Health Status and Self-Assessment of Health Condition, and the Relation to Health Services Utilization
Status: Completed | Type: Observational
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Collaborators: University of Haifa (Other)
Responsible Party: Sponsor
Other Study IDs: NHR-0049-14
Record Dates: First submitted 2016-05-02; First posted 2016-05-09 (Estimated); Last update posted 2016-05-09 (Estimated); Status verified 2016-05

CONDITIONS: Sf12-v2 Questionaire
Keywords: Self-assessment of health, Sf12-v2

STUDY DESIGN:
Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Sf12-v2 — structured questioner Sf-12v2, developed by Ware.et al (Ware, Kosinski, Turner-Bowker & Gandeck, 2002).

SUMMARY:
This study aims to examine the relation between health status and self-assessment of health condition, their relation to healthcare services utilization, and also to identify the profile of those who assess their health condition as mediocre to poor in general population and according to nationality.

DETAILED DESCRIPTION:
Background:

The World Health Organization defines "health" as a state of physical, mental and social well-being of an individual, and not just the absence of disease or illness. Health self-assessment is almost never present in medical and clinical models, which define "health" as the absence of physical disease. On the one hand, some say that there is a correlation between these definitions, and others argue that self-assessment of health is not always consistent with the clinical health status evaluation. Few studies have examined the relationship between self-assessment and health status among residents of the State of Israel in general and among the population residing in the Galilee and Western Galilee area in particular. The studies presented contradictory findings about the health perception among Jewish and Arab population. There are about 600,000 residents in Western Galilee from various population sectors, including Jews, Arabs, Druze and others. This composition of population pretty much reflects the general composition of population in the Galilee area.

Study objective:

This study aims to examine the relation between health status and self-assessment of health condition, their relation to healthcare services utilization, and also to identify the profile of those who assess their health condition as mediocre to poor in general population and according to nationality.

Methods:

A cross-sectional study was conducted among 250 visitors aged 18 and above of outpatient clinics in the Galilee Medical Center (former Western Galilee Hospital): opthalmology, dental, otolaryngology (ENT) and orthopedic. The target population group for this study is adult residents of the Western Galilee area. The sampling is random. For the aims of the survey five sampling days were selected in each of the four outpatient clinics. On each of the sampling days all visitors of different outpatient clinics were offered to complete a self-administered structured questionnaire adapted specifically for the study.

ELIGIBILITY:
Inclusion Criteria:

* Adult residents of the Western Galilee area

Exclusion Criteria:

* Non literate visitors

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Visitors at the outpatient clinics in the Galilee Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2014-09; Primary Completion 2014-10 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
A questionnaire on the self-assessment of one's health condition reflecting the physical condition and the illness status | 10 minutes

SECONDARY OUTCOMES:
A questionnaire used to correlate between illness status and health services utilization | 10 minutes
A questionnaire on the self-assessment of good health condition compared between Jews and Arabs. | 10 minutes

IPD SHARING:
Plan to Share IPD: No